CLINICAL TRIAL: NCT02694991
Title: Osteopathic Manipulative Treatment Efficacy in Sternal Pain Management After Heart Surgery
Brief Title: Osteopathic Manipulative Treatment Efficacy in Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001-2013
Record Dates: First submitted 2016-02-19; First posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Surgery; Pain
Keywords: surgery; outcome; pain; osteopathic manipulative treatment
MeSH Terms: conditions — Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OMT Group (Experimental): Osteopathic Manipulative Treatment 15 minutes once a day for 8 days
  Interventions: Other: Osteopathic Manipulative Treatment
- Control Group (No Intervention): No intervention, only usual care

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment — The thoracic wall is gently manipulated in conscious subjects in a supine position in order to facilitate greater diaphragmatic excursion. The thorax is palpated by applying a low pressure load directly on the skin in the direction of resistance, without any sliding over the skin or forcing of the subcutaneous tissue until it begins to yield and there is a sensation of softening. Sterile procedures are used when touching the patients near the surgical site. The treatment consists of a fixed and preordained sequence of three sessions, beginning with the costal arch on the diaphragm and then moving to the sternal area and, finally, the region of the thoracic outlet. The first two phases are performed from the right side, and the third from the head of the bed.
  Other Names: OMT
  Arms: OMT Group

SUMMARY:
Effectively controlling sternal pain during cardiac rehabilitation after heart surgery is very important as it reduces the risk of postoperative complications.

However, the contraindications and side effects of analgesic drugs may induce physicians to use them so cautiously that pain may actually be under-treated.

The aim of this open label, controlled study is to assess whether osteopathic manipulative treatment (OMT) can contribute to pain relief and improve rehabilitation outcomes.

DETAILED DESCRIPTION:
The currently predominant means of controlling postoperative pain is the peri-operative administration of opioid or non-opioid (acetaminophen) analgesics, alone or in combination, and non-steroidal anti-inflammatory drugs (NSAIDs). However, anti-inflammatory drugs are contraindicated for many patients because they may impair renal function, interact with platelet aggregation, and increase the risk of gastrointestinal damage and bleeding. The spectrum of available options is narrow.

Osteopathic manipulative Treatment (OMT) intervenes in the process that transforms nociceptive information into the subjective experience and it may be useful.

It has been found to be effective in controlling pain after abdominal surgery, it has a beneficial effect on patients recovering coronary artery by-pass surgery and also improves cardiac function The aim of this study was to assess whether complementary OMT is an effective means of reducing post-surgical sternal pain and improving rib cage mobility after heart surgery involving sternotomy, and to investigate its advantages during in-patient rehabilitation in terms of functional recovery, and perceived anxiety and depression.

This open, randomised, semi-blinded, controlled trial involves inclusion of 80 adult patients of both genders consecutively admitted as in-patients to cardiac rehabilitation unit after undergoing elective coronary artery by-pass grafting (CABG), valve replacement or repair and/or ascending aorta surgery with sternotomy, and capable of voluntarily providing their written informed consent. The patients are divided in 2 groups, the intervention group receiving OMT and the control group. Both groups are following the same rehabilitation programme and receiving usual care.

All of the subjects taking part in the study are receiving standard care in accordance with the international guidelines for in-patient cardiac rehabilitation; the only experimental intervention is the addition of OMT

ELIGIBILITY:
Inclusion Criteria:

* Recent artery bypass grafting (CABG)
* Recent valve replacement or repair
* Recent ascending aorta surgery

Exclusion Criteria:

* Heart surgery using mini-thoracotomy.
* Heart transplantation
* Implant of a ventricular assistance device
* Diabetes mellitus
* Rheumatoid arthritis
* Autoimmune diseases
* Altered cognitive capacities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-09; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Pain intensity relief | 21 days
  Pain intensity measured with visual analogic scale (VAS)

SECONDARY OUTCOMES:
Functional capacity improvement | 21 days
  Distance in meters walked in six minutes
Respiratory function | 21 days
  Inspiratory volume variation measured as mL of air inspired
Hospitalization length | 21 days
  Number of days of hospitalisation
Anxiety and Depression | 21 days
  Hospital Anxiety and Depression Scale (HADS) score
Analgesic drug consumption. | 21 days
  Number of analgesic drug doses taken

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Mocarelli, Prof, Study Chair — Fondazione Don C. Gnocchi
Locations (1):
- Fondazione Don C. Gnocchi ; Istituto S. Maria Nascente IRCCS, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
to upload the data base file of all results of the present trial